CLINICAL TRIAL: NCT01519063
Title: Glutamate-opioid Interactions in Alcohol Drinking Behaviors
Brief Title: Naltrexone and Memantine Effects on Alcohol Drinking Behaviors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 1005006779; P50AA012870 (NIH)
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Alcohol Drinking
Keywords: Alcohol; Drinking; Drinkers; Alcohol Drinking; Memantine; Naltrexone; Alcohol Dependence; Alcohol Abuse; Alcohol-Related Disorders; Ethanol; Alcoholism
MeSH Terms: conditions — Alcohol Drinking; Alcoholism; Alcohol-Related Disorders | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone and memantine (Experimental): Treatment with Naltrexone and memantine first
  Interventions: Drug: Naltrexone and memantine first; Drug: Naltrexone and Placebo first
- Naltrexone and Placebo (Placebo Comparator): Treatment with naltrexone and placebo first
  Interventions: Drug: Naltrexone and memantine first; Drug: Naltrexone and Placebo first

INTERVENTIONS:
Drug: Naltrexone and memantine first — Naltrexone 50mg memantine 20mg
  Other Names: memantine's brand name is Namenda; naltrexone's brand name is Revia
Drug: Naltrexone and Placebo first — Naltrexone 50 mg Placebo
  Other Names: naltrexone's brand name is Revia

SUMMARY:
The purpose of this study is to evaluate the combined effects of the study medications naltrexone and memantine on alcohol drinking behaviors.

DETAILED DESCRIPTION:
Participants will be randomized to receive a combination of naltrexone/memantine over a one week period and then participate in a laboratory session. During this session, participants are given an initial drink of alcohol followed by the choice to drink up to 12 more drinks over a three-hour period. These medications are hypothesized to reduce craving and number of drinks consumed prior to and after exposure to the initial drink of alcohol and during the three hour drinking period.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-55
* Able to read English at 6th grade level or higher and to complete study evaluations
* Regular alcohol drinker

Exclusion Criteria:

* Individuals who are seeking alcohol treatment
* Medical conditions that would contraindicate the use of study medication
* Regular use of other substances

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, Ph.D., Principal Investigator — Yale University
Locations (1):
- Sac, Cmhc, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants enrolled was 75. However, 19 people did not start medication due to ineligibility or drop out, leaving 56 total participants.
Groups:
- Naltrexone and Memantine First: Patients received Naltrexone and Memantine first in this arm.
- Naltrexone and Placebo First: Patients received Naltrexone and Placebo first in this arm.
Period: Overall Study
Arm/Group | Naltrexone and Memantine First | Naltrexone and Placebo First
Started | 26 | 30
Completed | 19 | 25
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Naltrexone and Memantine First: Patients in this arm received Naltrexone and Memantine first.
- Naltrexone and Placebo First: Patients in this arm received Naltrexone and Placebo first.
- Total: Total of all reporting groups
Arm/Group | Naltrexone and Memantine First | Naltrexone and Placebo First | Total
Number analyzed (Participants) | 26 | 30 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (8.5) | 33 (9.3) | 33 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 15 | 18 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Number of Caucasian and Non-Caucasian participants
  Participants
    Caucasian | 16 | 20 | 36
    Non-Caucasian | 10 | 10 | 20
Total number of drinks over past 90 days [Mean (Standard Deviation); unit: drinks] — Timeline Followback (TLFB; Sobell & Sobell, 1996)
  drinks | 166 (63) | 165 (1) | 165 (72)
Drinks per drinking day in past 90 days [Mean (Standard Deviation); unit: drinks] | 7.2 (2.5) | 7.2 (2.9) | 7.2 (2.7)
Percent of drinking days over past 90 days [Mean (Standard Deviation); unit: percent of days] | 78 (16) | 75 (17) | 76 (16)

OUTCOME MEASURES:

1. Primary Outcome: Number of Drinks Consumed at Lab Session (Day 7)
Description: Number of drinks consumed during the lab session (Day 7) after taking study medication, ranging from 0-12.
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: drinks
Groups:
- Naltrexone and Memantine: Treatment with Naltrexone and memantine
  Naltrexone and memantine: Naltrexone 50mg memantine 20mg
- Naltrexone and Placebo: Treatment with naltrexone and placebo
  Naltrexone and Placebo: Naltrexone 50 mg Placebo
Arm/Group | Naltrexone and Memantine | Naltrexone and Placebo
Number analyzed (Participants) | 47 | 46
drinks | 4.11 (4.19) | 5.02 (4.32)

2. Primary Outcome: Craving AUC: Adlib Drinking Phase
Description: Craving for alcohol based on Alcohol Urge Questionnaire (AUQ, Bohn et al., 1995), which is an 8 item measurement of self-reported alcohol urges that has been shown to be strongly related to alcohol dependence severity. Each item is scored from 1 (strongly disagree) to 7 (strongly agree), with a higher score indicating higher craving. Assessed multiple times, starting at 50 minutes after priming drink until 230 minutes after priming drink. Higher craving scores (ranging from 0-56) are indicated by larger log-transformed AUC.
Time Frame: 50-230 minutes after the priming drink during lab session
Measure: Mean (Standard Deviation); unit: log (units on a scale * minutes)
Arm/Group | Naltrexone and Memantine | Naltrexone and Placebo
Number analyzed (Participants) | 47 | 46
log (units on a scale * minutes) | 7.62 (.54) | 7.75 (.55)

3. Primary Outcome: Stimulation Response to Alcohol at Lab Session
Description: Brief Biphasic Alcohol Effects Scale-Stimulation subscale (BAES; Martin et al., 1993), measuring stimulation effects of alcohol. Seven items ranging from 0 (not at all) to extremely (10) with higher measurements indicating higher stimulation. Assessed multiple times, starting at 50 minutes after priming drink until 230 minutes after priming drink. Higher stimulation scores (ranging from 0-70) are indicated by larger log-transformed AUC.
Time Frame: 50-230 minutes after the priming drink during lab session
Measure: Mean (Standard Deviation); unit: log (units on a scale *minutes)
Arm/Group | Naltrexone and Memantine | Naltrexone and Placebo
Number analyzed (Participants) | 47 | 46
log (units on a scale *minutes) | 4.78 (3.51) | 4.93 (3.45)

4. Primary Outcome: Sedation Response to Alcohol at Lab Session
Description: Brief Biphasic Alcohol Effects Scale-Sedation subscale (BAES; Martin et al., 1993), measuring sedation effects of alcohol. The seven items included on the sedation subscale range from 1 (not at all) to extremely (10) with higher measurements indicating higher sedation. Assessed multiple times, starting at 50 minutes after priming drink until 230 minutes after priming drink. Area Under the Curve was used to calculate the final score reported for the BAES.
  As a single summary measure, AUC, was calculated for BAES outcomes based on scores recorded at numerous time points throughout the adlib drinking session The calculation was based on the trapezoidal methods using times 50, 90, 110, 150, 170, 210, and 230 . Based on the distribution, each AUC was log-transformed. Higher AUC levels correspond to greater levels of sedation.
Time Frame: 50-230 minutes after the priming drink during lab session
Measure: Mean (Standard Deviation); unit: log (units on a scale *minutes)
Arm/Group | Naltrexone and Memantine | Naltrexone and Placebo
Number analyzed (Participants) | 47 | 46
log (units on a scale *minutes) | 5.42 (2.97) | 5.34 (3.08)

5. Primary Outcome: Craving AUC: Priming Dose Phase
Description: Craving for alcohol based on Alcohol Urge Questionnaire (AUQ, Bohn et al., 1995), which is an 8 item measurement of self-reported alcohol urges that has been shown to be strongly related to alcohol dependence severity. Each item is scored from 1 (strongly disagree) to 7 (strongly agree), with a higher score indicating higher craving. Craving for alcohol based on Alcohol Urge Questionnaire is calculated using Area Under the Curve (AUC). A single summary measure, AUC was calculated for AUQ outcomes based on scores recorded at numerous time points throughout the priming drink session. The calculation was based on the trapezoidal methods using times -20, 10, 20, 30, 40, 50 minutes before/after priming drink. Based on the distribution, each AUC was log-transformed. Higher AUC levels correspond to greater alcohol urge.
Time Frame: 0-50 minutes after the priming drink
Measure: Mean (Standard Deviation); unit: log (units on a scale *minutes)
Arm/Group | Naltrexone and Memantine | Naltrexone and Placebo
Number analyzed (Participants) | 47 | 46
log (units on a scale *minutes) | 6.81 (.55) | 6.84 (.57)

6. Primary Outcome: Sedation Response to Alcohol: Priming Dose Phase
Description: Brief Biphasic Alcohol Effects Scale-Sedation subscale, measuring sedation effects of alcohol with higher measurements indicating higher sedation. Brief Biphasic Alcohol Effects Scale-Stimulation subscale (BAES; Martin et al., 1993), measuring stimulation effects of alcohol. Seven items ranging from 0 (not at all) to extremely (10) with higher measurements indicating higher stimulation. The subscale total range is 0-70, these scores are logged transformed.
Time Frame: 0-50 minutes after priming drink
Measure: Mean (Standard Deviation); unit: log (units on a scale)
Arm/Group | Naltrexone and Memantine | Naltrexone and Placebo
Number analyzed (Participants) | 47 | 46
log (units on a scale) | 3.87 (2.49) | 3.76 (2.34)

7. Primary Outcome: Stimulation Response to Alcohol: Priming Dose Phase
Description: Brief Biphasic Alcohol Effects Scale-Stimulation subscale, measuring stimulation effects of alcohol with higher measurements indicating higher stimulation. Brief Biphasic Alcohol Effects Scale-Stimulation subscale (BAES; Martin et al., 1993), measuring stimulation effects of alcohol. Seven items ranging from 0 (not at all) to extremely (10) with higher measurements indicating higher stimulation. The subscale total range is 0-70, these scores are logged transformed.
Time Frame: 0-50 minutes after priming drink
Measure: Mean (Standard Deviation); unit: log (units on a scale)
Arm/Group | Naltrexone and Memantine | Naltrexone and Placebo
Number analyzed (Participants) | 47 | 46
log (units on a scale) | 3.20 (2.84) | 3.43 (2.71)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at baseline and during the 7 days of medication, as well as at the one week follow up
Arm/Group | Naltrexone and Memantine | Naltrexone and Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/46
Other Adverse Events (participants affected / at risk) | 3/47 | 3/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone and Memantine (N=47) | Naltrexone and Placebo (N=46)
Nausea (Gastrointestinal disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT01519063/Prot_SAP_000.pdf